CLINICAL TRIAL: NCT00399776
Title: Bone Mineral Content and Bone Metabolism in Adolescents on Antipsychotic Therapy
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sriram Ramaswamy, M.D., Creighton University
Other Study IDs: 06-14216
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Adolescent Depression
Keywords: bone mineral; antipsychotic therapy; bone mineral accrual; bone mineral content
MeSH Terms: interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Adolescents taking haloperidol, risperidone, or olanzapine
  Interventions: Radiation: Bone Density Test
- Group B: Healthy adolescents
  Interventions: Radiation: Bone Density Test

INTERVENTIONS:
Radiation: Bone Density Test — Evaluating bone mineral content and bone metabolism in adolescents on antipsychotic therapy compared to healthy adolescents

SUMMARY:
We hypothesize that antipsychotic induced hyperprolactinemia can decrease bone mineral accrual and decrease bone mineral content (BMC) in adolescents on antipsychotic therapy.

Specifics Aims

1. To determine if antipsychotic therapy leads to decreased bone mineral accrual and decreased bone mineral content in a group of adolescents on antipsychotic therapy by comparing them to an ethnicity, gender and pubertal stage matched control group.
2. To determine the relationship between serum concentrations of prolactin, sex steroids and bone turnover markers in adolescents on antipsychotic therapy and an ethnicity, gender and pubertal stage matched control group.

DETAILED DESCRIPTION:
Recent studies have shown an increase in antipsychotic prescriptions among children and adolescents. Virtually all pediatric use of antipsychotics is "off-label," meaning without a Food and Drug Administration indication. To make matters worse, pediatric antipsychotic usage can lead to serious side effects like movement disorders and metabolic disturbances. Hence, it is concerning that despite the virtual absence of long term efficacy and safety data, the widespread use of antipsychotics in children and adolescents continues. One important adverse effects of antipsychotic therapy is hyperprolactinemia. Prolactin is a hormone secreted by the central nervous system. The main action of prolactin in females is the induction and maintenance of lactation. The main action of prolactin in females is the induction and maintenance of lactation. Antipsychotic therapy has shown to raise prolactin levels both, in the adult and pediatric population. Sustained hyperprolactinemia can cause a number of endocrinological abnormalities leading to a hypogonadal state and eventually bone demineralization and osteoporosis. There is evidence linking pediatric prolactinomas to decreased bone density. Also, adult studies suggest that the high rates of osteoporosis in schizophrenia may result from hypogonadism secondary to antipsychotic induced hyperprolactinemia. Our concern is that the sequela of antipsychotic induced hyperprolactinemia in children and adolescents, has received little attention, despite the important implications for bone health. This topic is especially important because peak bone mass is achieved during adolescence and is a key determinant of the lifetime risk of osteoporosis.

We hypothesize that antipsychotic induced hyperprolactinemia can interrupt bone mineral accrual and reduce bone mineral content in adolescents on antipsychotic therapy. We plan to measure bone mineral content and peripheral markers of bone metabolism in adolescents on antipsychotic therapy and compare them with ethnicity, gender and pubertal stage matched controls. We also plan to measure serum levels of prolactin and other hormonal measures such as: estradiol, progesterone, testosterone, follicle stimulating hormone, luteinizing hormone and thyroid function tests in both the groups. Statistical analysis will be performed to compare bone mineral content between the study and control groups. Additionally, the association between the hormonal measures and bone mineral content will be determined.

Osteoporosis is a major public health problem. In the United States today, 10 million individuals already have osteoporosis, and 18 million more have low bone mass, placing them at an increased risk for this disorder. Optimization of bone health is a process that must occur throughout the lifespan and factors that influence bone health at all ages are essential to prevent osteoporosis and its devastating consequences. To date, there are no published studies, examining the association between antipsychotic induced hyperprolactinemia and bone mineral content (BMC) and/or risk of osteoporosis in children or adolescents. Although there have been reports of antipsychotic induced hyperprolactinemia in both prepubertal and postpubertal children, it has been suggested that post pubertal children may be at a higher risk of decreased BMC. Thus, we plan to initially study the effects on adolescents. Potential implications of our research findings include: providing recommendations for preventing, diagnosing and monitoring bone mineral content/density during pediatric antipsychotic therapy. Since this is an unexplored area, yet very crucial field, findings from our study can be expected to have ramifications for clinical practice within one to two years of project completion.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent females and males with antipsychotic exposure equivalent to at least 100 chlorpromazine equivalents for a minimum of one year.
2. Age between 10 and 17 years of age
3. Within 10th and 90th percentile for height and weight -

Exclusion Criteria:

1. Pregnant
2. Chronic illness such as asthma, inflammatory bowel disease, rheumatoid disorders or cystic fibrosis.
3. On chronic systemic steroid therapy for the past 12 months
4. For subjects with hypothyroidism and on thyroid replacement therapy, TSH level will be obtained to determine eligibility.
5. Menstrual irregularities secondary to excessive physical activity.
6. History of anorexia nervosa and/or bulimia nervosa.
7. Subjects on hormonal contraception. -

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited from within the clinic as well as community psychiatrists
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Antipsychotic induced hyperprolactinemia can decrease bone mineral accrual | This is a 2 visit study

SECONDARY OUTCOMES:
Determine relationship between serum concentrations of prolactin, sex steroids and bone turnover markers in adolescents on antipsychotic therapy | This is a 2 visit study

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry Research Center, Omaha, Nebraska, United States